CLINICAL TRIAL: NCT01758588
Title: Phase II Randomized Controlled Trial of Pegylated Interferon Alpha-2b in Early Primary Myelofibrosis
Brief Title: Pegylated Interferon Alpha-2b in Early Primary Myelofibrosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was suspended due to insufficient subject accrual.
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1202012178
Record Dates: First submitted 2012-12-24; First posted 2013-01-01 (Estimated); Results first posted 2018-07-24 (Actual); Last update posted 2018-07-24 (Actual); Status verified 2018-06

CONDITIONS: Myelofibrosis
Keywords: Primary myelofibrosis; PMF
MeSH Terms: conditions — Primary Myelofibrosis | interventions — peginterferon alfa-2a; peginterferon alfa-2b; Interferon-alpha

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Observation arm (No Intervention): Subjects will be monitored closely for disease progression, however will receive no intervention.
- Peginterferon alfa-2a (Experimental): Peginterferon alfa-2a will be administered at a dose of 50 micrograms once a week for up to 3 years.
  Interventions: Drug: Peginterferon alfa-2a

INTERVENTIONS:
Drug: Peginterferon alfa-2a — 50 mcg subcutaneous injection once per week
  Other Names: PEGINTRON, Interferon alfa, IFNα-2b
  Arms: Peginterferon alfa-2a

SUMMARY:
The purpose of this study is to look at the effectiveness of giving patients who have been newly diagnosed with untreated early stage primary myelofibrosis (PMF) a study drug called PEGINTRON (also known as pegylated interferon alfa 2b). This intervention will be compared to the widely employed "watch and wait" (best supportive care) approach for early stage PMF, in which patients are followed closely and treatment initiated only if the disease progresses.

DETAILED DESCRIPTION:
Subjects will be randomized into one of the study groups: one in which subjects get treated with PEGINTRON and the other in which subjects are closely followed and get best supportive care until disease progression (the presently accepted standard approach for early disease). Subjects on the observation arm will be carefully monitored for clinical or laboratory progression of disease during scheduled study visits. However, they will not be treated with an active drug like Interferon alfa or others such as Hydroxyurea, Revlimid, Thalidomide, Pomalidomide, and the newly approved JAK2 (Janus Kinase 2) inhibitor Ruxolitinib (Jakafi). If their disease progresses, they will be eligible for cross-over into the treatment arm with PEGINTRON. Subjects randomized to the treatment arm will receive PEGINTRON once weekly.

ELIGIBILITY:
Inclusion Criteria:

- Patients must meet laboratory, and bone marrow histological criteria for primary myelofibrosis as defined by World Health Organization (WHO) diagnostic criteria as follows:

WHO diagnostic criteria for PMF Proposed Criteria for PMF Major Criteria

1. Presence of megakaryocyte proliferation and atypia, usually accompanied by either reticulin and/or collagen fibrosis, or, in the absence of significant reticulin fibrosis, the megakaryocyte changes must be accompanied by an increased bone marrow cellularity characterized by granulocytic proliferation and often decreased erythropoiesis (ie. prefibrotic cellular-phase disease)
2. Not meeting WHO criteria for Polycythemia Vera (PV), Chronic Myeloid Leukemia (CML), Myledysplastic Syndrome (MDS), or other myeloid neoplasm
3. Demonstration of JAK2617V>F or other clonal marker (e.g. MPL515W>L/K), or in the absence of a clonal marker, no evidence of bone marrow fibrosis due to underlying inflammatory or other neoplastic disease

Minor Criteria

1. Leukoerythroblastosis
2. increase in serum Lactase Dehydrogenase (LDH)
3. Anemia
4. Palpable splenomegaly

   * Patients must have Low or Intermediate 1 stage of disease as defined by International Working Group (IWG) risk stratification of primary myelofibrosis in the dynamic international prognostic scoring system (DIPSS). In addition, they must show some active hematopoiesis with a cellularity of at least 15%, irrespective of the degree of reticulin and/or collagen fibrosis as defined by Manoharan criteria.
   * Patients should NOT have had prior therapy for primary myelofibrosis. This includes treatment with cytoreductive drugs (Hydroxyurea), immunomodulatory drugs (thalidomide, lenalidomide, pomalidomide), JAK2 inhibitors, or other therapies specifically for myelofibrosis. If they received these classes of drugs for indications other than PMF, treatment should be discontinued at least 6 weeks prior to randomization.
   * Eastern Cooperative Oncology Group (ECOG) performance status < 2
   * Patients must have normal organ and marrow function as defined below:

     * White blood cell (WBC) ≥ 3,000/microL
     * Absolute Neutrophil Count (ANC) ≥ 1,500/microL
     * Platelets ≥ 100,000//microL
     * Total bilirubin within normal limits
     * Aspartate aminotransferase - serum glutamic oxaloacetic transaminase (AST(SGOT)) and alanine aminotransferase - serum glutamic pyruvic transaminase (ALT(SGPT)) less than or equal to 2.5 X upper limit of normal
     * Creatinine Clearance ≥ 50 ml/min
   * The effects of peg-IFNα-2b on the developing human fetus at the recommended therapeutic dose are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
   * Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria

* Patients who have had chemotherapy or radiotherapy within 6 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 6 weeks earlier.
* Patients with Intermediate 2 or High risk stage of disease as defined by International Working Group (IWG) risk stratification of primary myelofibrosis in the dynamic international prognostic scoring system (DIPSS) and/or bone marrow biopsy showing less than 15% cellularity in the presence +2 or more reticulin fibrosis (by Manoharan criteria), collagen fibrosis, or osteosclerosis.
* Patients may not be receiving any other investigational agents.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to peg-IFNα-2b
* Other Exclusion Criteria

  * Female patients who are pregnant or breast feeding
  * History of depression or active treatment for depression
  * History of non-compliance to medical regimens
  * History of autoimmune diseases
  * History of hypothyroidism or hyperthyroidism
  * Clinical evidence of neuropathy
* Uncontrolled illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant and lactating women are excluded from the study because the risks to an unborn fetus or potential risks in nursing infants are unknown.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-01; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard T Silver, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (2):
- United States (2):
  - Emory University Hospital, Atlanta, Georgia
  - Weill Medial College of Cornell Universiy, New York, New York

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients were randomized to either the treatment arm or the control arm of the study with a 2:1 allocation ratio. 8 patients were enrolled. No patients crossed over from observation to treatment.
Groups:
- Treatment Arm: 50mcg peginterferon alfa-2b subcutaneously per week
- Observation Arm: Patients were observed and did not receive treatment.
Period: Overall Study
Arm/Group | Treatment Arm | Observation Arm
Started | 5 | 3
Completed | 5 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment Arm: Patients treated with 50mcg of peginterferon alfa-2b subcutaneously per week.
- Observation Arm: Patients who did not receive treatment and were observed only.
- Total: Total of all reporting groups
Arm/Group | Treatment Arm | Observation Arm | Total
Number analyzed (Participants) | 5 | 3 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 3
  >=65 years | 4 | 1 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.9 (6.2) | 69.1 (5.5) | 69.9 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 3 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States: Weill Cornell Medicine | 4 | 2 | 6
  United States: Emory University | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Clinical Improvement
Description: Clinical improvement (CI) Requires one of the following in the absence of both disease progression (as outlined below) and Complete Response (CR)/Partial Response (PR) assignment (CI response is validated only if it lasts for no fewer than 8 weeks) i. A minimum 20-g/L increase in hemoglobin level or becoming transfusion independent (applicable only for patients with baseline hemoglobin level of less than 100 g/L).
  ii. Either a minimum 50% reduction in palpable splenomegaly of a spleen that is at least 10 cm at baseline or a spleen that is palpable at more than 5 cm at baseline becomes not palpable.
  iii. A minimum 100% increase in platelet count and an absolute platelet count of at least 50 000 109/L (applicable only for patients with baseline platelet count below 50 109/L).
  iv. A minimum 100% increase in Absolute Neutrophil Count (ANC) and an ANC of at least 0.5 109/L (applicable only for patients with baseline absolute neutrophil count below 1 109/L).
Time Frame: One year
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm | Observation Arm
Number analyzed (Participants) | 5 | 3
Participants
  Achieved Clinical Improvement (CI) | 1 | 0
  Did not achieve Clinical Improvement (CI) | 2 | 2
  Not evaluable | 2 | 1
Statistical Analysis 1: Comparison: Treatment Arm; Test type: Other; A statistical comparison and analysis of the clinical improvement (CI) proportions cannot be made because the sample size (n=5 in treatment arm, n=3 in observation arm) is too small

2. Secondary Outcome: Progression Free Survival
Description: Progression free survival is the measure of subject survival in the absence of disease progression. Disease progression is defined as progression to the next higher International Working Group-Myeloproliferative Neoplasms Research and Treatment (IWG-MRT) Dynamic International Prognostic Scoring System (DIPSS) stage from diagnosis. The IWG-MRT DIPSS stratifies primary myelofibrosis (PMF) into four risk categories (low, intermediate 1, intermediate 2, and high risk), based on 5 clinical factors; Age>65, Hemoglobin <10gm/dL, white blood cell (WBC)>25,000/uL, peripheral blasts>1%, and constitutional symptoms.
  Progression free survival will be assessed at 21 weeks from time of study entry.
Time Frame: Week 21
Population: Analysis population includes subjects who were evaluable at 21 weeks from time of study entry.
Measure: Count of Participants; unit: Participants
Groups:
- Treatment Arm: Subjects treated with 50mcg of peginterferon alfa-2b subcutaneously per week.
- Observation Arm: Patients were not treated and observed only.
Arm/Group | Treatment Arm | Observation Arm
Number analyzed (Participants) | 4 | 3
Participants
  Disease did not progress | 2 | 3
  Disease progressed | 2 | 0

3. Secondary Outcome: Overall Survival
Description: Overall survival measures subject survival regardless of disease progression.
  Overall survival will be assessed at 21 weeks from time of study entry.
Time Frame: Week 21
Population: Due to early termination of the trial, there is not enough data to evaluate overall survival.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm | Observation Arm
Number analyzed (Participants) | 4 | 3
Participants
  Not deceased | 4 | 3
  Deceased | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the date that the first patient was consented until study termination.
Description: The definitions of adverse event and/or serious adverse event, used to collect adverse event information, do not differ from the clinicaltrials.gov definitions.
Groups:
- Observation Arm: Patients on the non-interventional arm.
Arm/Group | Treatment Arm | Observation Arm
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/3
Serious Adverse Events (participants affected / at risk) | 2/5 | 0/3
Other Adverse Events (participants affected / at risk) | 1/5 | 0/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=5) | Observation Arm (N=3)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=5) | Observation Arm (N=3)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to early termination of the trial, there is not enough data to evaluate All-Cause Mortality. Therefore, it is reported that 0 subjects were affected out of 8 subjects at risk.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-10-30): https://cdn.clinicaltrials.gov/large-docs/88/NCT01758588/Prot_SAP_000.pdf